CLINICAL TRIAL: NCT00525993
Title: Efficacy and Safety of the Non-Steroidal Anti-Inflammatory Drug Etoricoxib in the Treatment of Acute Ankle Sprain in Sports: A Randomized Double-Blind Comparative Study Among 2 Treatments in the Acute Phase
Brief Title: Efficacy and Safety of Etoricoxib in Acute Ankle Sprain: A Double-Blind Comparative Study Among 2 Treatments Protocols
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Núcleo de Estudos em Esportes e Ortopedia, Brazil (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Rogerio Teixeira da Silva, NEO - Núcleo de Estudos em Esportes e Ortopedia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NeoBrazil_EtoricoxibAnkle2007
Record Dates: First submitted 2007-09-04; First posted 2007-09-06 (Estimated); Last update posted 2008-10-21 (Estimated); Status verified 2008-10

CONDITIONS: Sprains and Strains; Contusions
Keywords: sports; ankle; sprain; etoricoxib; antiinflammatory; treatment outcome
MeSH Terms: conditions — Sprains and Strains; Contusions | interventions — Etoricoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: etoricoxib 60mg daily for 14 days
- B (Active Comparator)
  Interventions: Drug: etoricoxib 90mg 14 days

INTERVENTIONS:
Drug: etoricoxib 90mg 14 days — each patient in this group will receive 90mg once daily, for the 14 days treatment.
  Arms: B
Drug: etoricoxib 60mg daily for 14 days — Patients in this group will receive 60mg of the drug, daily
  Arms: A

SUMMARY:
The investigators will study 2 doses of etoricoxib to prove that 60 mg once daily will be non-inferior to etoricoxib 90mg daily (for 14 days) in the treatment of acute ankle sprain in sports. The investigators objective is to discuss the point that the investigators will follow the minimal dose that is effective for the treatment of this acute condition in orthopedic.

DETAILED DESCRIPTION:
Study Objectives Primary

* To compare the efficacy of those 2 treatment doses in patients with acute ankle sprain in sports Secondary
* To compare the overall safety and tolerability of etoricoxib 60 mg and 90mg in patients with acute ankle sprain in sports

Hypothesis

* The efficacy of etoricoxib 60 mg once daily will be non-inferior to etoricoxib 90mg daily for 14 days in the treatment of acute ankle sprain in sports.
* The 60 mg dose of etoricoxib will have similarity in reducing the pain and will be more effective in decreasing the degree of edema, with most patients experiencing remission, which allows resumption of regular sporting activities after the end of the entire treatment.
* Both doses will be generally well tolerated and gastrointestinal intolerance will not be seen.

Background and Significance of the Selected Topic Etoricoxib is a cyclo-oxygenase (COX)-2-selective NSAID with a higher COX-1 to COX-2 selectivity ratio than the other COX-2-selective NSAIDs rofecoxib, valdecoxib or celecoxib. In patients with rheumatoid arthritis, improvements in tender and swollen joint counts and patient and investigator global assessment of disease activity were significantly greater in etoricoxib than in placebo recipients in two studies. Etoricoxib was also significantly more effective than naproxen in one of these studies. In patients with osteoarthritis of the hip or knee, etoricoxib was significantly more effective than placebo and had similar efficacy to naproxen with regards to improvements in pain and physical function scores and patient global assessment of disease status scores in two studies. Etoricoxib had similar efficacy to diclofenac in patients with osteoarthritis of the knee. Single-dose etoricoxib relieved pain in patients with postoperative dental pain in two studies. Similar scores assessing total pain relief over 8 hours (TOPAR8) were reported in etoricoxib and naproxen sodium or ibuprofen recipients, and higher TOPAR8 scores were reported with etoricoxib than with paracetamol (acetaminophen)/codeine. Pain relief was significantly better with etoricoxib than placebo in two studies in patients with chronic low back pain. Etoricoxib had similar efficacy to indomethacin in a study in patients with acute gout, and single-dose etoricoxib had similar efficacy to naproxen sodium in a study in women with primary dysmenorrhoea. Compared with non-COX-selective NSAIDs, etoricoxib was associated with significantly fewer upper gastrointestinal (GI) perforations, ulcers or bleeds, and was significantly less likely to result in treatment discontinuation because of NSAID-type GI symptoms or any GI symptoms.

There are a significant number of studies showing efficacy and superior GI tolerability profile of etoricoxib in chronic pathologies as mentioned above. However among acute pain pathologies there are a number of specific diagnosis that may be better explored. A very common diagnosis that causes acute pain are traumatic sport-related lesions of soft tissues (sprains, tendinitis, bursitis). One of the most common diagnosis is the acute ankle sprain, and many patients after an acute injury use the medication to control the pain and decrease the amount of edema.

Etoricoxib has been approved for acute pain in the dosage of 90 mg and it has been routinely prescribed for soft tissues inflammatory conditions, as acute gout. Otherway, we have some clinical cases that can lead to a longer period of pain, usually up to 2 weeks. As we know, when we have to use the medication for more than one week we have to decrease the dosage, and in some cases if you use a high dose it can lead to a persistent edema in the ankle joint. Therefore a study comparing etoricoxib 90 mg versus 60 mg in acute ankle sprain sport-related lesion is justified. As we know today, our efforts have to focus on usign the smallest dose to reach the best clinical results of a specific medication.

Study Design

* Study Type This will be a pilot study, randomized, single center, double-blind, parallel-group study to compare the efficacy and tolerability of etoricoxib 90 mg versus 60 mg in patients with acute ankle sprain.
* Sample Size The study will include 50 patients. One primary investigator (Rogerio Teixeira da Silva, MD, PhD) will coordinate the project.
* Study Medication and Flowchart

A total of 50 patients will be recruited to a randomized double-blind 14 days treatment study to evaluate the efficacy and the tolerability of oral etoricoxib 90mg daily in comparison with etoricoxib 60 mg/day in a 1:1 proportion.

• Study Procedures

Visit 1 / day 0 Screening: IC, Incl/excl criteria, MH, VS, PE, local injury exam, Lab tests: hemogram, biochemistry,, B-HCG (women), Hemoccult. Assessment of pain and pain during mobilization by VAS. Assessment of pain during motion against resistance, functional impairment, measurement of the edema (volumetric measurement) / Ultrasound examination of the ankle

Visit 2 / day 1 (may be allowed to perform with visit 1 if all lab tests are available).

Randomization: after complying with IC and all incl/excl criteria, 1 dose assisted. PE, local injury exam. Assessment of pain and pain during mobilization by VAS. Assessment of pain during motion against resistance, functional impairment.

Visit 3 / day 8 Evaluation for Adverse Experiences. VS, PE, local injury exam. Assessment of pain and pain during mobilization by VAS. Assessment of pain during motion against resistance, functional impairment and global assessment of efficacy and tolerability., measurement of the edema (volumetric measurement)

Visit 4 / day 15 End of treatment. Evaluation for Adverse Experiences, VS, PE, local injury exam, hemoccult. Lab tests: hemogram, biochemistry, B-HCG (women), Hemoccult. Assessment of pain and pain during mobilization by VAS. Assessment of pain during motion against resistance, functional impairment and global assessment of efficacy and tolerability. measurement of the edema (volumetric measurement)

Phone Contact / Day 45 After 4 weeks of completion of treatment, there will be a phone contact to assess resumption of regular sporting activities and adverse experiences in this period.

Efficacy Measures / endpoints of interest Primary • The main efficacy criterion will be the reduction of pain during active mobilization measured using a visual analogue scale VAS at day 8,. We will measure the normal movements of the joints (flexion and extension, abduction and adduction, external and internal rotation). Also we will evaluate the volumetric measurement of the ankle and foot, at day 1 and day 8.

Secondary

* The secondary efficacy criteria will be pain during motion against resistance, functional impairment and global assessment of efficacy by either patient and investigator, measured at Day 15. It will be measures by the VAS and also using the volumetric measurement.
* Tolerability will be assessed by the frequency of adverse experiences and global assessment of efficacy by either patient and investigator.

Statistics In this study we will include a total of 50 patients presenting acute ankle sprain occurred in sport, treat them with either oral etoricoxib (120 mg/day or 60 mg/day) for 14 days, under double-blind conditions, and verify efficacy and safety post-treatment accordingly.

Pain evaluation will be performed through a visual analog scale (VAS), ranging from 0 until 10, and median differences of one point in the VAS will be considered as significant. Based upon works using such scale, it was verified that the standard deviation within VAS is, in average, of 1.2 point.

According to methodology presented by Fisher & Belle (1993), the following table presents the sample estimation for different significances and study power:

Confidence Power Number necessary per group (ni) for 1-point difference in VAS

(1 - α) (1 - β) 0.95 0.95 37 0.95 0.90 30 0.95 0.80 23 0.90 0.95 31 0.90 0.90 25 0.90 0.80 18

Therefore, the number of patients for each study group would be 25 patients, with a confidence interval of 95% and study power of 90%. Considering the study as a pilot, we believe that this power is good. After this study, we can do another one to at least 74 patients to prove the more power of if.

ELIGIBILITY:
Inclusion Criteria:

* patients that suffered an ankle sprain in the last 12 hours and seek medical assistance

Exclusion Criteria:

* anterior history of trauma / fractures in the affected ankle
* history of hypertension / gastrointestinal problems
* patients that did not agree to sign the informed consent to participate in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-08 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Reduction of pain during active mobilization measured using a visual analogue scale VAS at day 8 | 8 days
Volumetric measurement of the ankle and foot | day 1 and day 8

SECONDARY OUTCOMES:
Pain during motion against resistance | day 15
Functional impairment and global assessment of efficacy by either patient and investigator | day 15
Tolerability will be assessed by the frequency of adverse experiences and global assessment of efficacy by either patient and investigator | day 15

CONTACTS AND LOCATIONS:
Overall Officials: Rogerio T Silva, MD, PhD, Principal Investigator — NEO - Orthopedic Sports Medicine Research Center; Lidia F Souza, PT, Study Director — NEO - Orthopedic Sports Medicine Research Center; Cristiano FS Laurino, MD, Study Director — NEO - Orthopedic Sports Medicine Research Center
Locations (1):
- NEO, São Paulo, São Paulo, Brazil